CLINICAL TRIAL: NCT01434810
Title: Treatment of Neonatal Jaundice With Filtered Sunlight Phototherapy: Safety and Efficacy in African Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1108M03601
Record Dates: First submitted 2011-08-30; First posted 2011-09-15 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Jaundice, Neonatal
Keywords: Hyperbilirubinemia, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Intervention Model Description: Non-inferiority trial comparing the two methods of phototherapy
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Filtered-sunlight phototherapy (Experimental): Infants will receive six hours per day of filtered-sunlight phototherapy for 1 to 10 days. The filtering will be done using window tinting film. Window tinting films by Solutia, Inc., and V-KOOL, Inc.
  Interventions: Device: Filtered-sunlight phototherapy
- Conventional phototherapy (Active Comparator): Infants will receive six hours per day of conventional phototherapy for 1 to 10 days.
  Interventions: Device: Conventional phototherapy

INTERVENTIONS:
Device: Filtered-sunlight phototherapy — Infants will receive six hours per day of filtered-sunlight phototherapy for 1 to 10 days. The filtering will be done using window tinting film. Window tinting films by Solutia, Inc., and V-KOOL, Inc.
  Arms: Filtered-sunlight phototherapy
Device: Conventional phototherapy — Infants will receive six hours per day of conventional phototherapy for 1 to 10 days.
  Arms: Conventional phototherapy

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of filtered sunlight phototherapy. Sunlight will be filtered by flexible (window-tinting) film. The subject population will be neonates born at Island Maternity Hospital, Lagos, Nigeria. The rationale for conducting the study is that in Nigeria, and other countries that may not have effective commercial light devices or have reliable access to electric power to operate them, filtered sunlight phototherapy might offer a safe and effective treatment for neonatal jaundice. Phase I of the study focused on the safety and efficacy of filtered sunlight phototherapy. Phase II of the study was a randomized controlled non-inferiority clinical trial comparing the efficacy of filtered sunlight phototherapy with conventional phototherapy.

DETAILED DESCRIPTION:
Numerous studies from resource-limited countries suggest that severe neonatal jaundice (NNJ) represents the largest unrecognized cause of neonatal morbidity and mortality in the world. Several studies from Africa rank jaundice as a leading cause of death in newborn nurseries. In Nigeria, Owa and Osinaike reported that jaundice (14%) was the second leading cause of death, while Ugwu et al, found that mortality from severe jaundice was comparable to birth asphyxia but greater than sepsis in neonates >24 hrs old to 7 days old. In Kenya, English et al reported NNJ as the third leading cause of both newborn admissions and deaths. Studies from Nigeria, Zimbabwe, Turkey, North Vietnam, Oman, and India listed acute bilirubin encephalopathy (ABE) and/or severe NNJ as a significant cause of morbidity, many of whom required exchange blood transfusion (EBT) in their nurseries. Unfortunately, phototherapy, as important as it is, may not be available to many infants with NNJ in these countries because of the lack of devices and/or of unreliable electrical power supply. Commercial phototherapy (PT) devices are expensive, often break down due to surges in electrical power, and are difficult to maintain due to unavailability of spare parts. Even where PT devices are available, most hospitals in these countries lack the resources to replace the fluorescent light bulbs at the recommended 2000-3000 hrs of use and simply leave ineffective tubes in place until they burn out. Moreover, very few hospitals have appropriate irradiance meters for monitoring the intensity of the blue light emitted by the lamps. In a recent study in Nigeria by Owa et al, none of the tested PT devices provided the level of irradiance required for intensive PT.

Often, the only treatment a healthcare provider can suggest to the parents/guardians of jaundiced infants is to place their babies in sunlight. However, this practice is unsuitable due to several safety concerns. For instance, exposure to ultraviolet (UV) light may cause sunburn, while infrared (IR) light may cause the body to overheat. Moreover, the infant may lose body heat from the uncovered skin during treatment, with potential for dehydration. A safer, yet practical and economical, solution is needed, providing the basis for our proposal of filtered sunlight PT.

The primary aims of this study were safety, efficacy and non-inferiority of filtered sunlight phototherapy compared to conventional phototherapy. Phase I of the study focused on the safety and efficacy of filtered sunlight phototherapy. Phase II focused on non-inferiority of efficacy as compared to conventional phototherapy while continuing to evaluate safety.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to participate in the study if all of the following conditions exist:

1. At time of birth, infant is > 35 weeks gestation (or > 2.2 kg if gestational age is not available
2. Infant is < 14 days old at the time of enrollment
3. At time of enrollment, infant has an elevated TcB defined as 3 mg/dL below the level recommended for high-risk infants per AAP guidelines or higher
4. Parent or guardian has given consent for the infant to participate

Exclusion Criteria:

Subjects will be excluded from participation in the study if any of the following conditions exist at the time of enrollment:

1. Infants with a condition requiring referral for treatment not available at the hospital study site and/or conventional phototherapy unit.
2. Infants with a life-expectancy of < 24 hours
3. Infants requiring oxygen therapy
4. Infants clinically dehydrated or sunburned
5. Infants with a temperature < 35.5 or > 38 degrees Centigrade
6. Infants with ABE on clinical exam
7. Infants meeting the criteria for EBT

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 447 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina M Slusher, MD, Principal Investigator — University of Minnesota
Locations (1):
- Island Maternity Hospital, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Slusher TM, Olusanya BO, Vreman HJ, Brearley AM, Vaucher YE, Lund TC, Wong RJ, Emokpae AA, Stevenson DK. A Randomized Trial of Phototherapy with Filtered Sunlight in African Neonates. N Engl J Med. 2015 Sep 17;373(12):1115-24. doi: 10.1056/NEJMoa1501074. PMID 26376136
- [Derived] Slusher TM, Olusanya BO, Vreman HJ, Wong RJ, Brearley AM, Vaucher YE, Stevenson DK. Treatment of neonatal jaundice with filtered sunlight in Nigerian neonates: study protocol of a non-inferiority, randomized controlled trial. Trials. 2013 Dec 28;14:446. doi: 10.1186/1745-6215-14-446. PMID 24373547

RESULTS

PARTICIPANT FLOW:
Groups:
- Filtered Sunlight Phototherapy: Window tinting film will be used.
  Window tinting film for filtered sunlight phototherapy: Six hours per day of filtered sunlight phototherapy for 1 to 10 days.
- Conventional Phototherapy: Infants will be randomized to conventional phototherapy (new arm)
  Conventional phototherapy: Conventional phototherapy unit will be used for infants randomized to this arm for 1 to 10 days.
Period: Overall Study
Arm/Group | Filtered Sunlight Phototherapy | Conventional Phototherapy
Started | 224 | 223
Completed | 201 | 213
Not Completed | 23 | 10
Not completed — Did not receive treatment | 11 | 3
Not completed — Missing data/received <5hr phototherapy | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Filtered Sunlight Phototherapy | Conventional Phototherapy | Total
Number analyzed (Participants) | 224 | 223 | 447
Age, Customized [Median (Inter-Quartile Range); unit: weeks]
  Est'd gestational age | 38 [38 to 39] | 38 [38 to 39] | 38 [38 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 103 | 205
  Male | 122 | 120 | 242

OUTCOME MEASURES:

1. Primary Outcome: Safety of Phototherapy
Description: For a given treatment day, the phototherapy treatment was deemed safe if that infant on that day did not have to be withdrawn from treatment due to hypo- or hyperthermia, sunburn or dehydration. Therefore safety is reported as a percentage of the total treatment days (i.e. number of safe treatment days divided by total number of treatment days).
Time Frame: Four to ten days
Population: Safety was assessed for all 593 days on which treatment was received, in all 433 participants who were treated.
Measure: Count of Units; unit: treatment days
Units Other Than Participants: treatment days
Arm/Group | Filtered Sunlight Phototherapy | Conventional Phototherapy
Number analyzed (Participants) | 213 | 220
Number analyzed (treatment days) | 268 | 325
treatment days | 268 | 325

2. Primary Outcome: Efficacy of Phototherapy
Description: For a given evaluable treatment day, the phototherapy treatment was deemed effective if that infant on that day had a decrease in serum bilirubin level or (if <72hrs old) an rate of increase of less than 0.2 mg/dL/h. Therefore efficacy is reported as a percentage of the evaluable treatment days (i.e. number of effective evaluable treatment days divided by total number of evaluable treatment days).
Time Frame: Four to ten days
Population: The efficacy analysis was carried out on the 561 treatment days which were evaluable (see flow chart).
Measure: Count of Units; unit: treatment days
Units Other Than Participants: treatment days
Arm/Group | Filtered Sunlight Phototherapy | Conventional Phototherapy
Number analyzed (Participants) | 201 | 213
Number analyzed (treatment days) | 250 | 311
treatment days | 232 | 280

3. Secondary Outcome: Number of Participants Requiring Exchange Blood Transfusion
Description: Exchange blood transfusion required to lower the bilirubin level. Serum bilirubin will be measured twice daily during filtered sunlight or conventional phototherapy exposure, for an expected average of four days, and a maximum of ten days.
Time Frame: Four to ten days
Population: The need for exchange blood transfusion was assessed on all 447 enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Filtered Sunlight Phototherapy | Conventional Phototherapy
Number analyzed (Participants) | 224 | 223
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Filtered Sunlight Phototherapy | Conventional Phototherapy
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/223
Other Adverse Events (participants affected / at risk) | 0/224 | 0/223

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No